CLINICAL TRIAL: NCT04856254
Title: Clinical and Ultrasound Score for Evaluation of Previous Cesarean Section Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Elsaeed Elgohary, Principal Investigator, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: previous cesarean section scar
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Previous Cesarean Section Scar
Keywords: Trial of labor after cesarean section(TOLAC)& vaginal birth after cesarean section (VBAC)

STUDY DESIGN:
Who Masked: Participant
Masking Description: The pregnant females will be classified according to clinical and ultrasound score as patient suitable to undergo trial of labor after CS [TOLAC] or not suitable for [TOLAC] so undergo from the beginning to elective repeated cesarean section.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Trial of labor after cesarean section — The pregnant females with history of previous cesarean section will be classified according to clinical and ultrasound score as patient suitable to undergo trial of labor after CS [TOLAC]or not suitable for [TOLAC] so undergo from the beginning to elective repeated cesarean section.
  Other Names: Elective repeated cesarean section

SUMMARY:
Cesarean delivery rates have increased dramatically worldwide. In the United States, cesarean section (CS) rates increased from 5% of all deliveries in 1970 to a high of 31.9% in 2016.Although efforts were made to reduce the number of CS, it failed to achieve the 15% rate recommended by the World Health Organization (WHO).Repeat CS is the most significant factor contributing to overall increased CS rates. The primary indication of repeat CS is a prior CS. The trial of labor after cesarean (TOLAC) is an attempt to reduce CS rates. Several national medical associations have provided practice guidelines for vaginal birth after cesarean section (VBAC), but these differ across countries.VBAC is relatively safe when compared with repeat CS.However, TOLAC rates have dropped significantly worldwide in recent years.

DETAILED DESCRIPTION:
Brief History taking include: age of patient, gravidity, parity, time interval between previous cesarean sections and current pregnancy, indication for the previous cesarean section, and fetal weight of previous delivery with special emphasis on menstrual history for proper dating and history of previous pregnancy to verify the inclusion or exclusion criteria.Physical examination include : General examination: for exclusion of presence of any medical disorders,Obstetric examination include: Fundal level to correlate with gestational age known by history, Umbilical grip to verify inclusion and exclusion criteria, Scar tenderness and shape in women who had undergone a previous cesarean section and investigations that will be performed including the following:basic routine antenatal investigations of pregnant women including blood group,Rhesus factor, complete blood count, blood sugar, and urine analysis. abdominal and transvaginal ultrasound will be performed for:a complete obstetric assessment at full term using TAS to confirm gestational age, fetal vitality, lie and presentation, amniotic fluid and placental position.Evaluation of the lower uterine segment using TVS, by measuring its thickness and identifying the echo structure for beinghomogenous or not . The LUS will be visualized in the sagittal section in the midline and lateral plane. The measurement will be obtained with the cursors at the urinary bladder wall- myometrium interface and the myometrium chorioamniotic membrane-amniotic fluid interface. Three layers can be identified by ultrasonography in a well-developed LUS in a midline section of sagittal view in a partially filled bladder. They are as follows from inside outwards:Chorioamniotic membrane with decidualized endometrium, a middle layer of myometrium and utero-vesical peritoneal reflection juxtaposed to muscularis and mucosa of the bladder.The lower uterine segment will be visualized in sagittal section in the midline.There after :150 patients will be evaluated using a measurement value of the clinical and ultrasound criteria and Follow up of all participants will be followed up till delivery, the mode of delivery either VBAC or elective repeated lower segment CS according to:History and clinical examination evaluation: Previous complicated CS or not, time interval between previous cesarean sections and current pregnancy(less than one year or more than one year),tender scar or not. US : TAS and TVS include: Lower uterine segment thickness , The echo structure of the lower uterine segment (Homogenous or nonHomogenous). For follow up of patient with previous CS include Initial evaluation: Each of the clinical and US parameters will be scored based on the sum of points is shown in table whatever to complete delivery by natural means or again by cesarean section.If the score is more than 7 out of 10 a vaginal birth will tried. On the other hand,Score 7 or less than 7 will be considered an indication to do repeated elective cesarean section.Careful follow up of patient during trial of labor after CS [TOLAC] for any possible symptoms and signs of uterine rupture that require immediate surgical intervention like : bleeding either intra abdominal or vaginal,cessation of uterine contraction,abnormal uterine contour,abdominal distention,shoulder tip pain,supraoubic pain,sudden severe abdominal pain may decrease after rupture,tender abdomen,rapid materinal pulse, low blood pressure,hypovolomic shock if rupture involve major blood vessels,no fetal presentation on vaginal examination,prolonged fetal bradycardia and absent fetal heart activity during continuous electronic heart rate monitoring.Careful examination of patient after vaginal delivery to detect any maternal complication by: local examination under anesthesia to ensure continuity of cesarean scar and ultrasound evaluation of scar.The parameters that are evaluated by clinical and ultrasound criteria Clinical and ultrasound criteria SCORE (2) SCORE (1)Tender scar Not tender (2) Tender (1)Previous complicated CS Not complicated (2) Complicated (1) ,Echo structure of the LUS Homogenous (2) Non homogenous (1)Lower uterine segment thickness More than or equal 3.65 mm(2) .more than 3mm to less than 3.65 mm(1)Pregnancy time interval after the CS More than 12 months(2) 12 months or less(1)Total Score (10) (5)

ELIGIBILITY:
Inclusion Criteria:

* Previous one cesarean section for non permenant indication.
* Pregnant women without any medical disorders.
* Gestational age: 36-40 weeks.
* Pregnant woman with singleton pregnancy.
* Clinically adequate pelvis.
* Normal ultrasonographic findings (gestational age, fetal structures and placental site).
* Cephalic vertex presentation.
* Patients not inlabour.

Exclusion Criteria:

* Previous repair of ruptured uterus.
* Women with history of long-term treatment for infertility.
* Multiple pregnancies.
* Previous operations in uterus rather than cesarean section.
* Polyhydramnios and Fetal macrosomia.
* Women with bad obstetric history (previous IUFD or difficult delivery).
* Disturbance of fetal heart rate (determined with the CTG).

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Novel score (Mosbah) score for evaluation of previous cesarean section scar | Baseline
  The aim of this study is to use a novel score (Mosbah score) for evaluation of previous cesarean section scar in pregnant women in order to select the best and most safe mode of delivery by using certain measurments based on clinical findings and ultrasound measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine - Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJK. Births in the United States, 2016. NCHS Data Brief. 2017 Sep;(287):1-8. PMID 29155684
- [Background] World Health Organization Human Reproduction Programme, 10 April 2015. WHO Statement on caesarean section rates. Reprod Health Matters. 2015 May;23(45):149-50. doi: 10.1016/j.rhm.2015.07.007. Epub 2015 Jul 27. No abstract available. PMID 26278843
- [Background] Cheng YW, Eden KB, Marshall N, Pereira L, Caughey AB, Guise JM. Delivery after prior cesarean: maternal morbidity and mortality. Clin Perinatol. 2011 Jun;38(2):297-309. doi: 10.1016/j.clp.2011.03.012. PMID 21645797
- [Background] Foureur M, Ryan CL, Nicholl M, Homer C. Inconsistent evidence: analysis of six national guidelines for vaginal birth after cesarean section. Birth. 2010 Mar;37(1):3-10. doi: 10.1111/j.1523-536X.2009.00372.x. PMID 20402716